CLINICAL TRIAL: NCT00184288
Title: Single Volume 1H MR Spectroscopy of Brain Metastases in Evaluation of Treatment Response.
Brief Title: Proton MR Spectroscopy of Brain Metastases in Evaluation of Treatment Response.
Status: Withdrawn | Type: Observational
Why Stopped: no patients recruited
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11184
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Melanoma
Keywords: Lipid; choline; metastasis; magnetic resonance spectroscopy; treatment response
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate the feasibility of in vivo single volume MR spectroscopy in evaluation of treatment response in patients with brain metastases, using 3T MR instrument. In order to optimize and avoid ineffective treatment of patients with brain metastases, in vivo MR spectroscopy can be an useful tool.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of brain metastases

Exclusion Criteria:

* children
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with brain metastases
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Lundgren, MD PhD, Study Director — Cancer clinic, St.Olavs Hospital Trondheim University Hospital
Locations (1):
- Norwegian University of Science and Technology, Faculty of Medicine, Trondheim, Norway